CLINICAL TRIAL: NCT04495452
Title: Precision Medicine in Anesthesia: Genetic Component in Opioid-induced Respiratory Depression
Brief Title: Precision Medicine in Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: Study initially halted due to the COVID pandemic because the research ventilator was repurposed for life saving efforts. Due to later clinical demands, the study was able to be restarted.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alethia Sellers, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300004738
Record Dates: First submitted 2020-04-27; First posted 2020-07-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample (about 10 mL) will be collected either during the IV line insertion or after fentanyl administration during the recovery period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Participants: We will be enrolling 200 participants, this will provide a large enough sampling to assure there are at least 25 patients with significant respiratory depression and 25 with insignificant respiratory depression.
  The genetic data from participants with the most respiratory depression defined as having a 20-40% decrease from initial respiratory parameters will be compared with genetic data from participants with the least respiratory depression defined as having no change or less than 10% decrease from initial respiratory parameters.
  Interventions: Drug: Fentanyl Drug Administration

INTERVENTIONS:
Drug: Fentanyl Drug Administration — Subjects will be given a standardized dose of fentanyl 2.5 mcg/kg estimated ideal body weight (males: ideal body weight = 50 kg + 2.3 kg for each inch over 5 feet. Females: Ideal body weight = 45.5 kg + 2.3 kg for each inch over 5 feet).

SUMMARY:
This study is designed to look at how often a decrease in the rate of breathing occurs after being given a routinely used intravenous (IV) pain medication. This pain medication (Fentanyl) is given in the research procedure room by the anesthesiologist. In addition to relieving pain, in some patients it has been observed that this medication may decrease the rate of breathing.

Different pieces of one's genetic makeup (also known as genes) can affect how well this medication relieves pain. The investigators do not know if these same genes influence how large the effect of the medication has on breathing rate. The purpose of this study is to determine if the presence or alteration of these same genes may be associated with a decrease in rate of breathing.

DETAILED DESCRIPTION:
Opioids are key analgesic drugs. Unfortunately, they have a high potential for abuse with potentially lethal consequences, more specifically death due to respiratory suppression. In both Canada and the US, the number of deaths from opioid overdose continues to rise at an alarming rate, far exceeding fatalities from motor vehicle accidents in Canada and becoming the number one cause of unintentional injury-related death in the US. In light of the opioid epidemic and CDC-scrutiny of opioid use, determining genetic profiles susceptible to respiratory depression could prove useful in further tailoring the treatment of pain both in the perioperative setting and in the chronic pain management setting.

The purpose of the proposed study is to evaluate for a genetic component of opioid-induced respiratory depression. Our overall study hypothesis is that genetic variation influences opioid-induced respiratory depression.

The primary aim of the study is to correlate an intravenous opioid bolus and genetic variations of opioid-related target genes. Secondary aims or outcomes are the determination of general variation in respiratory responses in response to a single intravenous fentanyl bolus. Other observed effects are age and gender related differences, the effect of a single fentanyl bolus on alertness, the incidence of emesis and opioid effects on micturition as determined by the modified Aldrete discharge criteria.

Based on existing work on genetic determinants of opioid receptor effects, we propose to correlate clinical parameters of respiratory depression (proportional reduction in respiratory minute ventilation) with the expression of single-nucleotide polymorphisms (SNPs) of genes related to opioid-induced analgesia. We propose to identify a subset of participants with the most significant respiratory depression and contrast those with participants that exhibit no respiratory effects. The blood samples from these two groups will be used to compare genetic variances of genes related to opioid-induced analgesia.

This will be a collaborative project between the clinical physicians and basic scientists in an effort to better characterize opioid-induced respiratory depression. We believe this work will be valuable as a means to prevent and treat opioid toxicity and guide development of safer approaches to opioid therapy and drug development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* older than 19
* able to follow the study instructions

Exclusion Criteria:

* Any medical condition that could affect study procedures or potentially put the subject at risk, in the opinion of the investigators
* age less than 18 or older than 40
* pregnancy
* obesity
* sleep apnea
* pulmonary problems such as moderate or severe bronchial asthma
* epilepsy
* chronic analgesic medication
* history of surgery for which details are unavailable
* allergy to fentanyl
* history of drug abuse
* positive urine test for illicit drugs
* female participants will be scheduled for a urine pregnancy test on the day of the procedure, prior to receiving study medication, only subjects with negative tests will continue

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will involve adult human volunteers, representative of the greater Alabama population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | From the time of administration of study medication to 10 minutes after study medication administration
  A decrease in breathing frequency as quantified by respiratory rate
Minute Ventilation | From the time of administration of study medication to 10 minutes after study medication administration
  A decrease in breathing as quantified by minute ventilation
Occlusion Pressure | From the time of administration of study medication to 10 minutes after study medication administration
  A measure of respiratory depression as quantified by occlusion pressure

CONTACTS AND LOCATIONS:
Overall Officials: Alethia Sellers, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No